CLINICAL TRIAL: NCT06132555
Title: Health Status and the Need for Social Return of Drug Abusers in Guangdong Province: a Secondary Data Analysis Study
Brief Title: Health Status and the Need for Social Return of Drug Abusers in Guangdong Province
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Wei XIA, PhD, Associate Professor, Sun Yat-sen University
Other Study IDs: WXIA-001
Record Dates: First submitted 2023-10-13; First posted 2023-11-15 (Actual); Last update posted 2023-11-15 (Actual); Status verified 2023-11

CONDITIONS: Drug Use
Keywords: drug abuser; health condition; social regression; secondary data analysis
MeSH Terms: conditions — Drug Misuse

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Drug abusers: Drug abusers who registered in any of the 80 streets and 40 towns selected according to the economic level and population distribution of each city and other reference standards have been included in the study. A total of 6906 valid questionnaires have been collected.
  The interviewees were selected from 5000 participants in the quantitative questionnaire. Priority is given to drug users who have abstained for more than three years, and all age groups under 30 years old, between 30 and 50 years old and over 50 years old are covered.
  Interventions: Other: Online questionnaire survey; Other: In-depth personal interview
- Drug rehabilitation institutions: The drug rehabilitation institutions included social work organization, compulsory detoxification center and rehabilitation center, which were selected according to the specific conditions of the selected cities, and the final number of participants was determined according to the personnel Settings of these institutions.
  Interventions: Other: Colloquia

INTERVENTIONS:
Other: Online questionnaire survey — The investigators have made an electronic questionnaire through the questionnaire star, and send the link or two-dimensional code of the electronic questionnaire to the subjects through WeChat or SMS to remind them to fill in the answer on the mobile phone or computer.
  The questionnaire consisted of four parts: (1) basic information of the interviewees, (2) drug abuse of the interviewees, (3) drug treatment interventions received by the interviewees, and (4) problems encountered by the interviewees when they return to society.
  Groups: Drug abusers
Other: In-depth personal interview — The in-depth personal interview was conducted in a semi-structured way. The outline of the interview was formulated from seven aspects: drug use history, drug abstinence history, relapse situation, living conditions, physical and mental health status, return to society status, and active drug abstinence willingness of the drug abstinence personnel. The aim was to understand the needs of drug addicts in terms of family relationship, peer relationship, history of drug use, history of drug withdrawal, employment, economy, social support network, psychology, and assistance.
  Groups: Drug abusers
Other: Colloquia — The colloquia were carried out in the form of group interviews, 1-2 people from each different institution were selected to participate, and the number of people in each colloquium was controlled to be between 6 and 12.
  The colloquia mainly focused on: ① The status quo of the implementation of the local drug drug treatment policy, ② the status quo of the compulsory isolation drug treatment work, ③ the status quo of the work of social workers for drug drug treatment, ④ the status quo of the work of community health centers, ⑤ the operation of various mechanisms in the work of various units, and ⑥ what content in the drug control work needs assistance from other departments and what external resources are needed.
  Groups: Drug rehabilitation institutions

SUMMARY:
This study intends to conduct a secondary analysis of the data from the investigation on the status quo of anti-drug rehabilitation work and management needs in Guangdong Province.

DETAILED DESCRIPTION:
The drug problem is a major problem that threatens individuals' physical and mental health, family happiness, national security, regional stability and world peace. In recent years, anti-drug departments in various regions of Guangdong Province have adhered to the arrangement and deployment of the National Anti-Drug Office, the provincial Party committee and the provincial government and the Party committee of the Public Security Department, focused on preventing the harm of synthetic drugs, improved the system, implemented responsibilities, and innovated methods, and constantly improved the anti-drug and drug rehabilitation work in Guangdong.

Nowadays, with the improvement of the level of social and economic development, the personnel structure and characteristics of drug abusers in Guangdong Province have undergone corresponding changes, and the effect of the existing control policies on drug abusers has also shown a weak stage, which needs to be adjusted and updated in time.

In this context, Guangdong Provincial Public Security Department has carried out research on anti-drug management countermeasures, and actively discussed the status quo, difficulties and reform direction of anti-drug management in the new era.

This study intends to conduct a secondary analysis based on the data obtained from the investigation and research on the status quo of drug control and detoxification work and management needs in Guangdong Province, aiming to describe the demographic and sociological characteristics of drug abusers in Guangdong Province, as well as their psychosocial experience of receiving interpretation intervention and the status quo of social regression needs. What's more, this study also devoted to forming a practical multi-department co-management model of community comprehensive management of drug addicts in Guangdong Province in the new era, to comprehensively improve the management level of drug abusers in Guangdong Province, serving grassroots communities, and build a harmonious society.

ELIGIBILITY:
Inclusion Criteria:

* Cities in Guangdong Province are selected according to the geographical distribution, development level, economic level and population distribution of the cities.
* Drug abusers who registered in any of a streets or townships of Guangdong Province would be selected.
* Drug abusers who have abstained for more than 3 years.
* All age groups under 30 years old, between 30 and 50 years old and over 50 years old were covered.

Exclusion Criteria:

* Eliminate more than 20 questions missed or not answered questionnaires.
* The questionnaires which be filled out by the same respondent repeatedly.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Drug abusers who registered in any of a streets or townships of Guangdong Province would be selected.
Sampling Method: Probability Sample
Enrollment: 7106 (Estimated)
Dates: Start 2023-11-15 (Estimated); Primary Completion 2024-07 (Estimated); Study Completion 2024-08 (Estimated)

PRIMARY OUTCOMES:
Health status | Baseline
  The main indicator of health status is the Brief Symptom Inventory-18 (BSI-18) scale, a simplified version of the commonly used psychological evaluation scale SCL-90, consisting of 18 items that are answered on a Likert scale of 0 to 4 points. A higher total score on the BSI-18 indicates a higher level of psychological distress for the respondent.

SECONDARY OUTCOMES:
Socio-demographic information of drug abusers | Baseline
  The socio-demographic data collected through the structural questionnaire includes gender, age, education level, income, family size and health status of drug abusers.
Withdrawal symptoms | Baseline
  The symptoms that the participants experienced during they quit the drugs. A checklist including 18 symptoms was used the measure the withdrawal symptoms with a Likert scale of 1 to 5 points. A higher score indicates more serious the participants experienced certain withdrawal symptoms.
Addiction treatment | Baseline
  The treatment that the participants ever received. A checklist including 4 common treatments used with a Likert scale of 0 to 4 points. A higher score indicates more effective in treating the drug abuse.
Barriers and support on returning to social | Baseline
  The barriers and support that the participants experienced when they tried to return to social. A checklist including 8 common barriers and 5 common support with a Likert scale of 1 to 4 points. A higher score indicates more serious or more necessary to the participants.

CONTACTS AND LOCATIONS:
Overall Officials: Wei Xia, PhD, Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Yes
The non-identified individual participant data will be shared after the outcomes have been published.
Supporting Information: SAP
Time Frame: After the publication of the study
Access Criteria: Researchers should contact the PI for approval of the study protocol.